CLINICAL TRIAL: NCT00099489
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Determine the Safety and Efficacy of AVONEX When Used in Subjects With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Brief Title: Safety and Efficacy of Avonex in Subjects With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec Medical Director
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-870
Record Dates: First submitted 2004-12-15; First posted 2004-12-16 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: Chronic Inflammatory Demyelinating Polyradiculoneuropathy; CIDP; IVIg; AVONEX
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Interferon beta-1a

INTERVENTIONS:
Drug: Interferon Beta-1a

SUMMARY:
The purpose of this study is to determine whether AVONEX (Interferon Beta-1a), when compared to placebo, reduces the total dose of IVIg that is administered after Visit 5 and through Visit 9 (Week 32, End of Study).

DETAILED DESCRIPTION:
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) is an acquired peripheral neuropathy of unknown origin. The etiology is not well understood but is presumed to be immunological. Evidence for this comes from observed similarities to Guillain-Barre syndrome and from the favorable response with immunomodulatory treatments.

CIDP is a peripheral nervous system demyelinating neuropathy that is sometimes a corollary disorder to the central nervous system demyelination of multiple sclerosis (MS. The precise mechanisms underlying the pathogenesis are uncertain, but a number of those mechanisms support a potential role for immunomodulatory treatments such as interferon beta (e.g., Biogen Idec Inc.'s AVONEX).

The rationale for the use of AVONEX in CIDP derives from observations on the pathogenesis of the condition and its similarities to MS, the mechanism of action of AVONEX, clinical trials that have been performed in CIDP that support a role for IFN-beta, and the unmet need that currently exists because of availability and safety issues with existing therapies.

This Phase 2b study is a dose-ranging study designed to provide scientific evidence regarding the safety and efficacy of AVONEX in CIDP. In addition, the study aims to demonstrate the responsiveness and clinical relevance of changes in the MRC sum score and ODSS in CIDP patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any testing under this protocol
* Must be between 18 and 75 years of age
* Have a diagnosis of CIDP as determined by a board-certified or board-eligible neurologist, or equivalent, for at least 6 months, including fulfilling modified INCAT neurophysiological criteria for CIDP,CIDP motor deficit responsive to IVIg and alternative EP data that justifies subject inclusion, and/or supportive pathologic or laboratory data that supports the diagnosis of CIDP
* Documentation in the medical record prior to screening that the CIDP had been associated with loss of muscle strength, such that the MRC sum score was less than or equal to 58.
* Documentation in the medical record that the patient benefited fom IVIg treatment (patient had a 2-point change or equivalent in 60-point MRC sum score)
* Tested for IgM monoclonal gammopathy and found to have tested negative for IgM monoclonal gammopathy or if positive for IgM monoclonal gammopathy, then are MAG antibody-negative and proven to be IVI g responsive per protocol.
* Must have been clinically stable while on a constant regimen of IVIg (every 2-weeks, 3-weeks, 4-weeks or 5-weeks) in the 3 months prior to screening.

Exclusion Criteria*:

* Associated systemic disorder that might cause neuropathy.
* History of, or abnormal laboratory results indicative of any significant major disease or known drug hypersensitivity that, in the opinion of the investigator, would preclude the administration if IFN-beta or participation in this study.
* Subjects with diabetes mellitus will not be eligible, unless they satisfy both of the following requirements: a) their diabetes is well-controlled, with no retinopathy or nephropathy, having been identified during the ongoing care of their diabetes; and b) they have a normal sensory nerve action potential (SNAP) amplitude recorded in the sural nerve on at least one side of the body identified during electrophysiology (EP) testing documented in their medical record.
* Abnormal screening or baseline blood tests that the investigator deems clinically significant
* History of a seizure disorder prior to baseline (Visit 1, Week 0).
* History of suicidal ideation within 3 months prior to Baseline Visit (Week 0) or an episode of severe depression within 3 months prior to Baseline Visit (Week 0).
* Pure motor syndrome fulfilling criteria for multifocal motor neuropathy with conduction block.
* Pure sensory CIDP, or any other variant of CIDP without motor involvement
* Serious local infection or systemic infection within the 6 months prior to Screening.
* Use of IFN-beta at any time, use of plasma exchange, plasmapheresis, or any other immunosuppressant (with the exception of oral or non-systemic corticosteroids) within 6 months prior to Screening.
* History of intolerance to acetaminophen (paracetamol), ibuprofen, naproxen, and/or aspirin that would preclude use of at least one of these during the study.
* For female subjects, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception, as defined by the Investigator, during the study.
* Female subjects considering becoming pregnant while in the study
* Female subjects who are currently pregnant or breast-feeding.

  * This list is not exhaustive and there may be additional exclusions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67
Dates: Start 2004-02; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for the efficacy analyses is the total IVIg dose (g/Kg) administered after Visit 5 and through Visit 9 (Week 32, End of Study).

SECONDARY OUTCOMES:
The time to disease progression.
Percentage reduction in IVIg dose (g/Kg).
The number of days between Visit 5 and either disease progression or Visit 9
(Week 32, End of Study).
The proportion of subjects with disease progression at Visit 9 (Week 32, End of Study).
The change in MRC sum score from baseline to the time of IVIg withdrawal.
Change from baseline to Visit 5 and to Visit 9 (Week 32, End of Study) in a composite score of maximal conduction velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Ropper, MD, Principal Investigator — Tufts University School of Medicine, St. Elizabeth's Medical Center; Kate Dawson, MD, Study Director — Biogen
Locations (20):
- United States (13):
  - Phoenix Neurological Associates, Ltd., Phoenix, Arizona
  - Neuromuscular Research Center, Scottsdale, Arizona
  - University of Florida, Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of Kansas, Kansas City, Kansas
  - Louisiana State University, New Orleans, Louisiana
  - Harvard University/MGH, Boston, Massachusetts
  - Tufts University/ St. Elizabeths, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Weill Medical College of Cornell University, New York, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Institute of Clinical Neurosciences, Sydney, New South Wales
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (2):
  - London Health Sciences Center, London, Ontario
  - Montreal Neurological Hospital, Montreal, Quebec
- Guy's Hospital/Dept. of Neuroimmunology, London, United Kingdom